CLINICAL TRIAL: NCT02284763
Title: Pharmacodynamic Modeling of the Effect of End-tidal Carbon Dioxide on Cerebral Oxygen Saturation in Beach Chair Position Under General Anesthesia
Brief Title: Modeling the Effect of EtCO2 on Cerebral Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2014-0688
Record Dates: First submitted 2014-10-20; First posted 2014-11-06 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Shoulder Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Change of EtCO2 (Experimental): Changes of rSO2 after adjustment of EtCO2 between 27-45 mmHg
  Interventions: Other: EtCO2

INTERVENTIONS:
Other: EtCO2 — Initial data collection during BCP was performed following three conditions were satisfied: after start of surgery; at least 15 min after BCP (for stabilization of MAP); after ventilation frequency was adjusted to produce EtCO2 of 27-29 mmHg with tidal volume of 8 ml/kg. Data was collected every 3 min after decreasing ventilation frequency by 1-2 breaths/min to increase EtCO2 until 42-45 mmHg. Once the value of EtCO2 42-45 mmHg was reached, ventilator frequency was increased in the same way to decrease EtCO2 until 27-29 mmHg. Fraction of inspired oxygen of 50% was maintained and end-tidal desflurane concentration was adjusted to achieve bispectral index values of 40-55 during data collection.

SUMMARY:
The aim of this study was to investigate the relationship between the end-tidal carbon dioxide (EtCO2) and cerebral oxygen saturation (rSO2) and to identify the covariates in the pharmacodynamic relationship between EtCO2 and rSO2.

DETAILED DESCRIPTION:
Even though mild hypercapnia in the beach chair position (BCP) under general anesthesia was effective in reducing cerebral desaturation, there is no comprehensive data with regard to the dose-effect relationship of EtCO2 on rSO2 in the BCP under general anesthesia. Pharmacodynamic modeling can be useful in describing this relationship in which concurrent mean arterial pressure changes and disease state can be considered as covariates. Therefore, we investigated the relationship between the EtCO2 and rSO2 and identified the covariates in the pharmacodynamic relationship between EtCO2 and rSO2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years who were scheduled to elective arthroscopic shoulder surgery in BCP under general anesthesia

Exclusion Criteria:

* Previous cerebrovascular disease, orthostatic hypotension, and the American Society of Anesthesiologists physical status IV or V

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The parameters of indirect response model | 60 min
  fractional turnover rate (kout), baseline rSO2, baseline EtCO2, linear slope governing the relation between EtCO2 and rSO2
The factors that influence the model parameters | 60 min
  mean blood pressure, end-tidal desflurane concentration, age, sex, hypertention, diabetes mellitus, weight

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, MD, PhD, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea